CLINICAL TRIAL: NCT01265628
Title: Validation of the GATE Software for Static Visual Field Examinations
Brief Title: Validation of the GATE Software
Acronym: ValGATE
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Haag-Streit AG (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Prof. Dr. med. Ulrich Schiefer, University Hospital Tuebingen
Other Study IDs: HSC GATE Strategie; 161/2009BO2 (Other: Ethics Committee University Hospital Tübingen)
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Visual Field Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Glaucoma
  Interventions: Procedure: perimetry
- Retinitis pigmentosa (RP)
  Interventions: Procedure: perimetry
- Anterior Ischemic Optic Neuropathy (AION)
  Interventions: Procedure: perimetry

INTERVENTIONS:
Procedure: perimetry — automated static perimetry with adapted GATE strategy
  Other Names: Octopus 900

SUMMARY:
Comparison of the differential luminance sensitivity (DLS) values at each test point

ELIGIBILITY:
Inclusion Criteria:

* physical, intellectual and linguistic abilities, in order to understand the test requirements
* spherical ametropia max. ± 8 dpt, cylindrical ametropia max. ± 3 dpt
* distant visual acuity > 10/20
* isocoria, pupil diameter > 3 mm

Exclusion Criteria:

* pregnancy, nursing
* diabetic retinopathy
* asthma
* HIV+ or AIDS
* history of epilepsy or significant psychiatric disease
* medications known to effect visual field sensitivity
* acute ocular infections (e.g. keratitis, conjunctivitis, uveitis)
* severe dry eyes
* miotic drugs
* amblyopia
* squint
* nystagmus
* albinism
* keratoconus
* intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening
* history or presence of macular disease and / or macular edema
* relevant opacities of central refractive media (cornea, lens, vitreous body)
* ocular trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: selected from the eye hospital's database
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Validation of visual field data and comparison of the differential luminance sensitivity (DLS) values at each test point by applying two perimetric software versions. | up to 14 days
  each participant were examined 2 times at two seperate sessions within 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof.Dr.med., Principal Investigator — University of Tuebingen, Centre for Ophthalmology
Locations (1):
- Centre for Ophthalmology, Institute for Ophthalmic Research, Tübingen, Germany

REFERENCES:
- [Derived] Luithardt AF, Meisner C, Monhart M, Krapp E, Mast A, Schiefer U. Validation of a new static perimetric thresholding strategy (GATE). Br J Ophthalmol. 2015 Jan;99(1):11-5. doi: 10.1136/bjophthalmol-2013-304535. Epub 2014 Jul 22. PMID 25053761